CLINICAL TRIAL: NCT05726032
Title: Effects of Empagliflozin on Natriuresis and Volume Overload in Patients With Cirrhosis and Ascites
Brief Title: Empagliflozin in Patients With Cirrhosis and Ascites
Acronym: EMPA Liver
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000034606
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cirrhosis; Liver Failure
MeSH Terms: conditions — Fibrosis; Liver Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Proof of concept, randomized, cross over, phase II double-blind placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Active Comparator): Empagliflozin vs placebo for 14 days, followed by 14 day washout period, before crossing over to the alternate drug.
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Empagliflozin vs placebo for 14 days, followed by 14 day washout period, before crossing over to the alternate drug.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Participants will be randomized to Empagliflozin 10 mg or placebo for 14 days. A 14 day washout period follows and then participants is crossed over to the alternate treatment for 14 days.
  Arms: Empagliflozin
Drug: Matching Placebo — Participants will be randomized to Empagliflozin 10 mg or placebo for 14 days. A 14 day washout period follows and then participants is crossed over to the alternate treatment for 14 days.
  Arms: Placebo

SUMMARY:
A proof-of-concept placebo-controlled trial to explore the acute and 14-day effects of empagliflozin on natriuresis and total body water in patients with cirrhosis and ascites. We will additionally investigate its effect on neurohumoral activation, and renal hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cirrhosis and ascites on a stable dose of diuretics (spironolactone +/- loop-diuretics based on AASLD guidelines)10 and who do not require large volume paracenteses
2. eGFR >= 30mL/min/1.73 m2
3. >=18 years old

Exclusion Criteria:

1. Hospitalization due to a complication of cirrhosis in the previous 8 weeks (e.g. variceal hemorrhage, encephalopathy, acute kidney injury, spontaneous bacterial peritonitis)
2. Direct bilirubin >=3 mg/dL
3. Systolic blood pressure < 100 mmHg
4. Active malignancy including hepatocellular carcinoma undergoing treatment
5. History of bladder dysfunction, incontinence, pyelonephritis, urosepsis, or frequent urinary tract infections
6. Use of SGLT-2 inhibitors in the last 10 days, or previous use with intolerance
7. Type 1 diabetes
8. History of frequent hypoglycemic episodes
9. Use of a non-loop diuretic aside from aldosterone antagonists or amiloride as they are not standard of care in patients with cirrhosis and could potentially increase the risk of hypovolemia when combined with the standard treatment for ascites along with SGLT2 inhibitor.
10. Hepatic hydrothorax requiring thoracentesis in the prior 8 weeks
11. Hepatic encephalopathy grade II or greater at the time of enrollment
12. Patients who have had TIPS placed
13. Previous liver transplant
14. Participation in another trial with an investigational drug within the 30 days prior to informed consent
15. Pregnancy or breastfeeding
16. Inability to give written informed consent or follow study protocol (e.g. clinically-significant psychiatric, addictive, or neurological disease)
17. Change in diuretic dose in the prior 2 weeks
18. Patients with hospitalization for alcoholic hepatitis in the past 6 months
19. Significant worsening of creatinine (more than 50% increase) in the past 4 weeks
20. MELD-Na > or equal to 20
21. Hemoglobin <8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in FENa with administration of study drug (10 mg empagliflozin vs. identical placebo) | 14 days
  Change in fractional excretion of sodium with administration of study drug (10 mg empagliflozin vs. identical placebo)
Change in total body water (TBW) before and after a 14-day course of study drug | 14 days
  Change in total body water (TBW) before and after a 14-day course of study drug (10 mg/day empagliflozin vs. identical placebo)

SECONDARY OUTCOMES:
Change in renal blood flow before and after administration of study drug | Baseline to Hour 6
  Change in renal blood flow (RBF) as determined by PAH clearance, before and after the acute administration of study drug ((RPF assessed using ancillary protocol on page 31)
Change in plasma renin activity,total renin, aldosterone, norepinephrine and copeptin | 14 days
  Change in plasma renin activity (PRA), total renin, aldosterone, norepinephrine and copeptin before and after a 14-day course of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No